CLINICAL TRIAL: NCT03580811
Title: The Clinical Effect of Simultaneous Grafting With Implant Placement Comparing Soft Tissue Grafting Alone to Combined Hard and Soft Tissue Grafting
Brief Title: Clinical Effects of Hard and Soft Tissue Grafting With Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18.0470
Record Dates: First submitted 2018-06-13; First posted 2018-07-09 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Dental Implants
Keywords: Alloderm; Dental Implants; Alveolar bone grafting
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: two groups of 15 patients . One with soft tissue grafting and implant placement and other with soft and hard tissue grafting with implant placement.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dental Implant & ADMG (Active Comparator): Dental implant placed with simultaneous grafting using one layer of ADMG
  Interventions: Device: Dental Implant &ADMG
- Dental implant & ADMG & BDX (Experimental): Dental implant placed plus simultaneous grafting using ADMG with BDX
  Interventions: Device: Dental Implant &ADMG; Device: Dental implant & ADMG & BDX

INTERVENTIONS:
Device: Dental Implant &ADMG — A dental implant will be placed and the buccal soft tissue will be grafted using ADMG .
Device: Dental implant & ADMG & BDX — Dental Implant will be placed with ADMG that covers the BDX
  Arms: Dental implant & ADMG & BDX

SUMMARY:
The study will be done to see if Implant placement and simultaneous grafting using alloderm alone will result in the same facial ridge contour and soft tissue thickness as alloderm plus bovine derived xenograft. Is the facial soft tissue contour and thickness for alloderm plus bovine derived xenograft is significantly increased compared to alloderm alone.

DETAILED DESCRIPTION:
Thirty sequentially entered patients will have a dental implant placed in maxillary sites from 4 to 13. Any implant system is acceptable since the objective of the study is to evaluate soft tissue contour due to graft placement, not to evaluate the implant. Once selected for participation immediately prior to treatment, they are randomized for a treatment group by a coin toss. Fifteen patients will receive Alloderm alone (Positive Control Group) while another fifteen will receive Alloderm plus Bovine derived Xenograft (Test Group). The graft will be placed simultaneously with the dental implant. A blinded examiner Dr.Jodie Lusby will be used. Should the examiner become unblinded the subject will be excluded from the study. Means and standard deviations will be calculated for all parameters. A paired test will be used to evaluate the statistical significance of the differences between initial and final data. An unpaired t-test will be used to evaluate statistical differences between the test and control groups. A sample size of 12 will afford ≥ 80% statistical power to detect a difference of 0.4 mm soft tissue thickness between groups. P value will be set at p≤0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Have one edentulous site bordered by 2 teeth in maxillary sites from second premolar to second premolar (maxillary 4 to 13) to receive an implant with simultaneous grafting with an ADMG with or without BDX.
2. Healthy persons at least 18 years old.
3. Understands and has signed the informed consent.

Exclusion Criteria:

1. Patients with uncontrolled diabetes, immune disease, or any systemic disease that significantly affects the periodontium.
2. Previous head and neck radiation.
3. Patients who have taken oral bisphosphonates for > 3 years or any IV bisphosphonates.
4. Smokers (or other tobacco habits that might interfere with soft tissue healing).
5. Patients who need prophylactic antibiotics prior to dental procedures.
6. Patients with allergies to any medication or material used in the study, or that would adversely affect study procedures.
7. Chemotherapy in the previous 12 months.
8. Psychological problems that would interfere with treatment.
9. Pregnant subjects will be excluded due to risk of miscarriage
10. Patients unable or unwilling to sign the informed consent.

    -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Buccal soft tissue contour around dental implant | 3 months
  Contour will be categorized as concave,flat or convex(subjective categories).

SECONDARY OUTCOMES:
Buccal soft tissue thickness around dental implants | 3 months
  The thickness will be measured with an endodontic file using a rubber stopper(objective measure of tissue thickness by penetrating tissue and measuring thickness in millimeters (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, MSD, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No